CLINICAL TRIAL: NCT02382198
Title: A Randomized, Placebo-controlled, 2-arm Parallel-group Superiority Phase II Study of GLYCOpyrrolate for Moderate-to-severe Sialorrhea in PARkinson's Disease
Brief Title: Study of Glycopyrrolate for Moderate-to-severe Sialorrhea in Parkinson's Disease
Acronym: GLYCOPAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OttawaHRI REB 2015-0043
Record Dates: First submitted 2015-01-21; First posted 2015-03-06 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Sialorrhea; Parkinson's Disease
Keywords: droooling, sialorrhea, parkinson's disease, parkinsons
MeSH Terms: conditions — Sialorrhea; Parkinson Disease | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Group (Active Comparator): This arm will receive the study drug glycopyrrolate.
  Interventions: Drug: Glycopyrrolate
- Placebo Group (Placebo Comparator): Control arm to receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glycopyrrolate — Drug to reduce drooling in patients with Parkinson's Decease.
  Arms: Active Group
Drug: Placebo
  Arms: Placebo Group

SUMMARY:
Sialorrhea is a frequently occurring problem with detrimental effect on quality of life in 25% of PD patients. Currently, there is no intervention approved for sialorrhea in Parkinsons and evidence is only available for a 30-day effect or less. We hypothesize that glycopyrrolate will have a lasting effect in the reduction of sialorrhea in PD patients.

DETAILED DESCRIPTION:
To assses if Glycopyrrolate has a long lasting effect on sialorrhea for patients with Parkinsons.

ELIGIBILITY:
Inclusion Criteria:

* PD as defined by United Kingdom PD Society Brain Bank criteria
* Moderate-to-severe sialorrhea defined by a score in the item 2.2 of the MDS-UPDRS greater than 2

Exclusion Criteria:

1. Other idiopathic parkinsonian syndromes, e.g., Progressive Supranuclear Palsy, Cortico-basal syndrome, or Multiple System Atrophy
2. Secondary parkinsonian syndromes (drug-induced, traumatic, encephalitic or vascular)
3. Change in antiparkinsonian medication one month prior to enrolment
4. Prior use of glycopyrrolate with or without known hypersensitivity will be considered an exclusion criterion, as it increases the risk of unblinding due to prior knowledge of potential side effects or therapeutic benefit
5. Change in the dose one month prior to enrolment of other anticholinergic agents or other drugs potentially affecting saliva production, such as tricyclic antidepressants, MAO-A inhibitors, neuroleptics (including clozapine and quetiapine more frequently used in PD) or hypnotics. These medication will remain in a constant dose throughout the trial;
6. Concomitant use of solid oral dosage forms of potassium chloride;
7. Pregnancy, breastfeeding, and premenopausal females or males not using adequate contraception; medically acceptable birth control methods for this study include: (1) Abstinence (no sexual intercourse); (2) Intrauterine device (IUD); (3) Diaphragm with spermicide; (4) Condom with spermicide; and (5) Oral contraceptives (birth control pills) + condom/diaphragm with spermicide.
8. Moderate-to-severe constipation in spite of optimal treatment (MDS-UPDRS, item 1.11>2);
9. Conditions that preclude anticholinergic therapy, e.g., documented history or symptoms suggestive of inflammatory bowel disease, glaucoma, myasthenia gravis, prostatic hypertrophy or obstructive urinary symptoms;
10. Conditions that can be exacerbated by anticholinergic effects of glycopyrrolate, e.g., documented history or symptoms suggestive of congestive heart failure, coronary heart disease, gastro-esophageal reflux disease or hyperthyroidism;
11. Uncontrolled arterial hypertension (TAS>140 mmHg or TAD>90 mmHg, using an electronic sphygmomanometer and standardized procedure16);
12. Tachyarrhythmia (interval RR <0.6 sec.);
13. TSH<0.4 mIU/L;
14. Liver dysfunction (AST, ALT, ALP >2xUpper Normal Limit);
15. Renal dysfunction (creatinine clearance <50 mL/min), as glycopyrrolate has predominant renal clearance;
16. Inability or unwillingness of subject or legal guardian/representative to give written informed consent;
17. Clinical significant lactose intolerance or known hypersensitivity to any of the study medication excipients
18. Participation in another investigational study at the time of recruitment or during the prior month.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mean sialorrhea related-disability at end of treatment (day 90) measured by the patient/caregiver-rated ROMP-saliva. | 90 days

SECONDARY OUTCOMES:
Mean score in sialorrhea severity at end of treatment (day 90) measured by the sialorrhea scoring scale | 90 days
Proportion of participants with a reduction of severity of sialorrhea in at least one point from baseline to end of treatment (day 90), measured by the MDS-UPDRS, item 2.2. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Mestre, MSc, MD, Principal Investigator — The Ottawa Hospital
Locations (2):
- Canada (2):
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided